CLINICAL TRIAL: NCT04512040
Title: Feasibility of At-Home Telehealth Yoga for Treating Chronic Pain
Brief Title: At-Home Telehealth Yoga for Treating Chronic Pain in People With Alzheimer's Disease and Their Caregiver's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Peter Bayley, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAY0006AGGAD; 3R34AT010364-02S1 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-13 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease; Musculoskeletal Pain; Chronic Pain
Keywords: Alzheimer Disease; yoga; telehealth; caregiver
MeSH Terms: conditions — Alzheimer Disease; Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned a treatment group for the duration of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Dyads AD patients and Caregivers (Experimental): Initially Yoga will be delivered in 1-on-1 format between the yoga therapist and the AD/caregiver dyad. Five outpatient adults, with chronic musculoskeletal pain and a diagnosis of mild AD and their Caregiver, will receive at-home teleyoga classes via video conferencing. Later, yoga will be delivered in a group format. Ten outpatient adults with chronic musculoskeletal pain and a diagnosis of mild AD and their Caregiver will receive group at-home teleyoga classes via video conferencing.
  Interventions: Behavioral: At-Home Yoga

INTERVENTIONS:
Behavioral: At-Home Yoga — At-home yoga practice over 12 weeks.

SUMMARY:
This feasibility study will evaluate yoga as a treatment for chronic pain in people living with Alzheimer's disease, and their Caregivers. The experimental treatment is yoga delivered via a tablet computer to participants at home ("teleyoga").

DETAILED DESCRIPTION:
The investigators will demonstrate the feasibility of conducting a trial involving teleyoga for people with Alzheimer's disease and their Caregivers. Participants with Alzheimer's disease and chronic pain (n=15) and their Caregivers (n=15) will all participate in teleyoga classes. Yoga classes will be given weekly for 12 weeks. At the end of treatment, participants will provide feedback by completing a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

AD PATIENTS

Inclusion Criteria for AD patients (As determined by):

* Diagnosis of probable Alzheimer's disease- Baseline
* Mini-Mental State Examination (MMSE) score 18-25 (Mild AD)(screening interview)
* ≥ 18 years old
* Has a primary care provider who can provide medical clearance for participation in the study
* Diagnosis of chronic musculoskeletal pain > 6 months
* Minimum pain intensity at screening visit: pain rated ≥4 on a 0-10 Numeric Rating Scale (NRS)
* Not begun new pain treatments or medications in the past month
* If on a psychotropic medication regimen: stable regimen for at least 4 weeks prior to entry to the study; willingness to remain on a stable regimen during the 12-week acute treatment phase
* English literacy
* Wireless internet connection at home (Screening interview)
* Has a caregiver who is willing to accompany AD patient for treatment, and who can receive yoga treatment at the same time as AD patient.

Exclusion Criteria for AD patients (As determined by):

* Participation in another concurrent clinical trial
* Back surgery within the last 12 months
* Back pain potentially attributed to a specific underlying cause, disease, or condition (VA EMR; screening interview)
* Baseline pain <4 or ≥9 on a 0-10 Numeric Rating Scale (NRS)

Inclusion Criteria for CAREGIVERS of AD patients (As determined by):

* Are caring for a patient diagnosed with AD who will practice yoga together with them
* Has a primary care provider who can provide medical clearance for participation in the study (Yoga Medical Clearance Form)
* Exclusion Criteria for Caregiver
* Participation in another concurrent clinical trial
* Attended or practiced yoga ≥ 1 x in the past 12 months
* Attended or practiced yoga ≥ 1 x in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bayley, PhD, Principal Investigator — PAVIR/VA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified electronic data sets of outcomes will be made available.
Supporting Information: SAP
Time Frame: End of treatment
Access Criteria: upon written request to the corresponding author of the manuscripts that are generated from this project

RESULTS

PARTICIPANT FLOW:
Groups:
- AD Patients; Caregivers: Yoga will be delivered in either a 1-on-1 format or a group format between the yoga therapist and the AD/caregiver dyad.
  Participants will receive at-home teleyoga classes via video conferencing.
Period: Overall Study
Arm/Group | AD Patients | Caregivers
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- AD Patients; Caregivers: Yoga will be delivered in 1-on-1 format between the yoga therapist and the AD/caregiver dyad.
  Participants will receive at-home teleyoga classes via video conferencing.
- Total: Total of all reporting groups
Arm/Group | AD Patients | Caregivers | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 1 caregiver did not provide their age at baseline
  Years
    number analyzed (Participants) | 15 | 14 | 29
    (all) | 73.33 (9.79) | 63.86 (9.31) | 68.60 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number of analyzed in rows differ from overall number due to no responses by some participants.
  Participants
    number analyzed (Participants) | 13 | 14 | 27
    Female | 10 | 10 | 20
    Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Attendance
Description: % of classes attended in 12 weeks of treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of classes attended
Arm/Group | AD Patients | Caregivers
Number analyzed (Participants) | 14 | 14
percentage of classes attended | 85.12 (15.75) | 86.31 (15.19)

2. Other Pre Specified Outcome: Treatment Satisfaction: Questionnaire
Description: Satisfaction of treatment was measured using the Multi-Dimensional Treatment Satisfaction Measure (MDTSM), which is composed of 33 questions that assess treatment process and outcome attributes.
  Each of the 33 questions is scored on a zero to 4 Likert rating scale with a score of zero indicating "not at all satisfied" and a score of 4 indicating "very satisfied". For each participant the mean score from all 33 ratings is calculated, which produces a score ranging from zero (not at all satisfied) to 4 (very satisfied). For the assessment of feasibility, we set the group mean target score on the MDTSM to ≥2, representing neutral or positive satisfaction.
Time Frame: immediately after the final treatment session (1 day)
Population: 1 dyad dropped out during intervention, 1 dyad lost to follow up after intervention (total of 13 dyads completed outcome measures)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AD Patients | Caregivers
Number analyzed (Participants) | 13 | 13
score on a scale | 3.01 (0.69) | 3.30 (0.63)

ADVERSE EVENTS:
Time Frame: baseline to end of treatment (12 weeks)
Arm/Group | AD Patients | Caregivers
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04512040/Prot_SAP_ICF_000.pdf